CLINICAL TRIAL: NCT04534400
Title: Automated Quantification of Radiologic Pulmonary Alteration During Acute Respiratory Failure: Application to the COVID-19 Pandemic
Brief Title: Automated Quantification of Radiologic Pulmonary Alteration During Acute Respiratory Failure
Acronym: QUANTICO-RETRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: VISIBLE PATIENT, E-MEDIA (Unknown)
Responsible Party: Sponsor
Other Study IDs: 7888
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: SARS-CoV-2 Infection; Respiratory Failure With Hypoxia
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with SARS-CoV-2 infection
  Interventions: Radiation: thoracic CT-scan
- Patients with Postoperative hypoxemic respiratory failure
  Interventions: Radiation: thoracic CT-scan

INTERVENTIONS:
Radiation: thoracic CT-scan — Automated measurement

SUMMARY:
Automated quantification of the pulmonary volume impaired during acute respiratory failure could be helpful to assess patient severity during COVID-19 infection or perioperative medicine, for example.

This study aim at assessing the correlation between the amount of radiologic pulmonary alteration and the clinical severity in two clinical situation :

1. SARS-CoV-2 infections
2. Postoperative hypoxemic acute respiratory failure

ELIGIBILITY:
Inclusion Criteria:

* patient with insurance covering
* patient admitted to the participating hospitals for SARS-CoV-2 infection or postoperative acute hypoxemic respiratory failure between 01/01/2019 and 05/11/2020

Exclusion Criteria:

- patient transferred to another hospital than the participating center during the 7 days following the CT scan

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients that underwent a thoracic CT-scan
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between altered pulmonary volume and ordinal severity scale | 2 days after CT scan

SECONDARY OUTCOMES:
Correlation between altered pulmonary volume and ordinal severity scale | 7 days after CT scan

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - HÔPITAUX UNIVERSITAIRES DE STRASBOURG, Hôpital de Hautepierre, Service de Réanimation Médicale, Strasbourg
  - Hôpitaux Universitaires de Nancy Service d'anesthésie réanimation Hôpital de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No